CLINICAL TRIAL: NCT05522790
Title: Impact of Iron Infusion in Anemic Patients on Their Postoperative Outcome After Colorectal Surgery
Acronym: IRON_PREHAB
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: IRON_PREHAB
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Anemia, Iron Deficiency; Colorectal Surgery
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2005, colorectal surgery in France represented nearly 40,000 procedures per year, of which 80% were scheduled and 70% were for carcinological purposes. Overall postoperative mortality was estimated at 3.4%, morbidity at 35% and average length of stay at 18 days. In addition, the number of newly diagnosed cases of colorectal cancer was 44,872 in 2017, making it the second leading cause of cancer in women and the third in men. The implementation of colorectal Enhanced Rehabilitation After Surgery (EARS) programs has resulted in a significant reduction in length of stay due to an approximately 50% decrease in postoperative complication rates and a faster return of patients to independence. However, despite the integration of RASC into routine practice, morbidity remains high with an estimated complication rate of 15-20%. The persistence of a high complication rate despite the rehabilitation measures can be explained in part by factors present preoperatively that impair postoperative recovery, such as the existence of comorbidities, low functional capacity, the presence of martial or nutritional deficiencies or glycemic imbalance. Links between the presence of these different "deficits", which may coexist, and postoperative morbidity and mortality have already been shown.

Anemia is common in preoperative colorectal surgery and affects approximately one in two patients with cancer. In case of preoperative anemia, the frequency of postoperative complications and the length of stay are increased. Under these conditions, preoperative correction of anemia could facilitate postoperative recovery and reduce the incidence of postoperative complications. In colorectal cancer, anemia is the consequence of an absolute martial deficiency due to iron losses from bleeding and a functional martial deficiency due to decreased availability of iron for erythropoiesis due to inflammation. Correction of preoperative anemia is usually based on 2 types of molecules: iron and erythropoiesis stimulating agents. Erythropoiesis-stimulating agents are not recommended to correct anemia in cancer patients not receiving chemotherapy. Iron can be given orally or intravenously. Intravenous administration is more effective than oral administration in patients with colorectal cancer to correct preoperative anemia. In patients undergoing colon cancer surgery outside of a RAAC program, preoperative iron infusion appears to decrease the incidence of postoperative complications, improve the quality of postoperative recovery, and reduce length of stay. These gains do not appear to be related to correction of preoperative anemia, since preoperative intravenous iron increases hemoglobin levels by only 0.8 g/dl, on average. And, insufficiently to reduce the rate of postoperative transfusion in abdominal or general surgery. Also, the benefits observed with preoperative iron infusion seem to be more related to the direct effects of iron on cardiac and skeletal muscle than by correction of anemia. Since 2016, all patients undergoing scheduled colorectal surgery at the Paris Saint Joseph Hospital Group benefit from the application of a RAAC program. If we do not take into account patients who die during hospitalization (≈ 2%) and patients transferred to Follow-up and Rehabilitation Care (SSR) (≈15%), the impact of the application of a RAAC program is easily measured with the length of stay. Indeed, reducing the frequency of postoperative complications and improving the speed of postoperative recovery translates into reduced lengths of stay. Today, the average length of stay for all patients undergoing colorectal surgery at Saint Joseph Hospital is 7.5 days. The length of stay is longer (8.7 days) in patients with anemia preoperatively compared to those without anemia (7 days). Since 2017, anemic patients scheduled for colorectal surgery, have received intravenous iron infusion preoperatively at Paris Saint Joseph Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age and older
* Patient operated on for colorectal surgery between January 1, 2017 and December 31, 2021
* Patient with preoperative anemia (12 g/dl for women, 13 g/dl for men)
* Patient hospitalized in conventional hospitalization

Exclusion Criteria:

* Patient undergoing emergency surgery
* Patient without preoperative hemoglobin measurements
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient opposing participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patient operated on for colorectal surgery between January 1, 2017 and December 31, 2021, with preoperative anemia (12 g/dl for women, 13 g/dl for men)
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Postoperative recovery speed | Month 1
  This ouctome corresponds to the postoperative length of stay, which corresponds to the difference between the date of discharge and the date of the operation.

SECONDARY OUTCOMES:
Rate of medical complications | Month 1
  This ouctome corresponds to the distribution of patients according to the severity of postoperative medical complications measured with the Clavien Dindo scale.
Rate of surgical complications | Month 1
  This ouctome corresponds to the distribution of patients according to the severity of postoperative surgical complications measured with the Clavien Dindo scale.
Rate of patients transfused | Month 1
  This ouctome corresponds to the percentage of patients transfused and number of red blood cells (RBCs) per patient transfused.
Postoperative hemoglobin level | Month 1
  This ouctome corresponds to the Postoperative hemoglobin level (nadir) corresponding to the lowest value measured postoperatively and before transfusion of packed red blood cells.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal ALFONSI, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Greco M, Capretti G, Beretta L, Gemma M, Pecorelli N, Braga M. Enhanced recovery program in colorectal surgery: a meta-analysis of randomized controlled trials. World J Surg. 2014 Jun;38(6):1531-41. doi: 10.1007/s00268-013-2416-8. PMID 24368573
- [Background] Munoz M, Laso-Morales MJ, Gomez-Ramirez S, Cadellas M, Nunez-Matas MJ, Garcia-Erce JA. Pre-operative haemoglobin levels and iron status in a large multicentre cohort of patients undergoing major elective surgery. Anaesthesia. 2017 Jul;72(7):826-834. doi: 10.1111/anae.13840. Epub 2017 Apr 6. PMID 28382661